CLINICAL TRIAL: NCT06044493
Title: A Multicenter, Randomization, Open-label Phase 4 Clinical Trial to Evaluate the Efficacy and Safety of MYREPTIC-N® or MY-REPT® in Stable Patients After Kidney Transplant Recipients
Brief Title: MYREPTIC-N® or MY-REPT® in Stable Patients After Kidney Transplant Recipients
Acronym: MyMy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B130_01KT2203
Record Dates: First submitted 2023-08-24; First posted 2023-09-21 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Kidney Transplant
Keywords: Kidney transplant; Mycophenolic acid
MeSH Terms: interventions — Mycophenolic Acid; Capsules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Myreptic-N Tablet (Experimental): Mycophenolate sodium
  Interventions: Drug: Myreptic-N Tablet
- Myrept Tablet/Capsule (Active Comparator): Mycophenolate mofetil
  Interventions: Drug: Mycophenolate mofetil Tablet/Capsule

INTERVENTIONS:
Drug: Myreptic-N Tablet — Up to 720mg BID(total 1440mg daily), PO - Check the blood concentration of Mycophenolate at each visit
  Other Names: Myreptic-N®
  Arms: Myreptic-N Tablet
Drug: Mycophenolate mofetil Tablet/Capsule — Up to 1g BID(total 2g daily), PO - Check the blood concentration of Mycophenolate at each visit
  Other Names: Myrept® Cap./Tab.
  Arms: Myrept Tablet/Capsule

SUMMARY:
The purpose of this study is to Evaluate the Efficacy and Safety of MYREPTIC-N® or MY-REPT® in Stable Patients after Kidney Transplant Recipients

DETAILED DESCRIPTION:
This study is a multi-center, Randomized, Open-label and phase IV clinical trial that evaluates the efficacy and safety of MYREPTIC-N® or MY-REPT® administration for 24 weeks in renal transplant patients combined Calcineurin inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Over 19 years old
2. Patients who at least 1 year after kidney transplant
3. serum creatinine ≤2.3 mg/dL
4. Patients on immunosuppressive maintenance therapy using combination of Calcineurin Inhibitor and Mycophenolate Mofetil after kidney transplantation

Exclusion Criteria:

1. Patients who had received treatment Acute rejection within 4 weeks
2. Patients who had discontinued corticosteroid within 4 weeks
3. At the time of Screening

   * Treatment with active liver disease or Liver function test(T-bilirubin, AST, ALT)is over 3 times than upper normal limit
   * WBC< 2,500/mm^3, or platelet < 75,000/mm^3, or ANC < 1,300/ mm^3
4. In investigator's judgement

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of composite efficacy failure | Until 24 weeks
  Composite efficacy failure include biopsy-confirmed acute rejection, graft loss, death, or follow-up failure

SECONDARY OUTCOMES:
Change in survey evaluation score [Gastrointestinal symptom rating scale(GSRS), EuroQol-5D(EQ-5D)] | Changes in scores from the baseline at week 24
  The GSRS consists of 15 questions, with a total score of 15 to 105, indicating that the higher the total score, the more severe the gastrointestinal symptoms.
  The EQ-5D evaluates quality of life and consists of 5 questions. Each question is evaluated in the range of 1 to 5. The score is calculated according to EQ-5D index. Calculated score is lower that means poor health.
Intra patient variability of mycophenolic acid | Until 24 weeks
  Measurement of blood levels of mycophenolic acid
Intra patient variability of calcineurin inhibitor | Until 24 weeks
  Measurement of blood levels of calcineurin inhibitor
Incidence of Virus infection | Until 24 weeks
  Frequency of incidence (BK Virus, CMV)
Incidence of biopsy-confirmed acute rejection | Until 24 weeks
  Frequency of incidence
Incidence of Graft loss | Until 24 weeks
  Frequency of incidence
Incidence of Death | Until 24 weeks
  Frequency of incidence

CONTACTS AND LOCATIONS:
Overall Officials: Jongwon Ha, MD, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea